CLINICAL TRIAL: NCT02301559
Title: The Influence of the Method Pilates in Life Quality, Intensity of Pain and Flexibility of Women With Primary Dysmenorrhea
Brief Title: The Influence of the Method Pilates in Women With Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual do PiauÍ (Other)
Responsible Party: Principal Investigator, Juliany Marques Abreu da Fonseca, academic physiotherapy, Universidade Estadual do PiauÍ
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04008402357J
Record Dates: First submitted 2014-11-16; First posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pilates Group (Experimental): Pilates Group, Pilates exercises, 20 sessions, lasting 40 minutes each, 3 times per week. Soil and ball exercises, with emphasis on the pelvic region. The program began with the work of breathing and postural correction, with warm-up exercises or preparatory, followed by the framework of classical movements of the method.
  Interventions: Behavioral: Pilates exercises

INTERVENTIONS:
Behavioral: Pilates exercises — Pilates exercises with emphasis on pelvic region

SUMMARY:
Primary dysmenorrhea is the result of hypercontractility and uterine vascular ischemia is the most common gynecologic complaints in young women. According to the intensity of symptoms may impair daily living, work and leisure activities. Pilates brings the concept of moving the body for the recovery, maintenance and promotion of health through exercises that stimulate circulation, improving physical conditioning, flexibility and proper postural alignment, and promote improvement in the levels of body awareness, coordination and muscle control. In this sense, the objective is to investigate the effects of pilates in the symptomatology of primary dysmenorrhea. This is a study to be developed with students of Physical Therapy from the State University of Piauí-UESPI presenting with primary dysmenorrhea compatible clinical picture. A questionnaire will be used for research. The students with the framework of dysmenorrhea that meet the inclusion criteria will be assessed for anthropometric parameters, pain, flexibility, indirect assessment of contraction of transversus abdominis and quality of life before and after the treatment protocol using the pilates method, often 3 weekly meetings, totaling 20 sessions.

DETAILED DESCRIPTION:
The objective is to investigate the effects of pilates in the symptomatology of primary dysmenorrhea. This is a study to be developed with students of Physical Therapy from the State University of Piauí-UESPI presenting with primary dysmenorrhea compatible clinical picture. A questionnaire will be used for research. The students with the framework of dysmenorrhea that meet the inclusion criteria will be assessed for anthropometric parameters, pain, flexibility, indirect assessment of contraction of transversus abdominis and quality of life before and after the treatment protocol using the pilates method, often 3 weekly meetings, totaling 20 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary
* Female
* 18-25 years old
* Enrolled in Physiotherapy course at the State University of Piauí- UESPI, with symptoms compatible with primary, nulliparous dysmenorrhoea, who have regular menstrual cycle and who agree to participate spontaneously in the research, by signing a term of informed consent (Appendix a) in accordance with Resolution 466/2012.
* Participation in the survey did not veto the use of analgesic or contraceptive by the participants.
* All are oriented to maintaining the habits of life - food, work and leisure activities, medications - during the exercises

Exclusion Criteria:

* Will not be included in the selected research volunteers that do not show symptoms and characteristics consistent with primary dysmenorrhoea according to the questionnaire, and those who accept not participate and / or not signing the consent form sample.
* As criteria for inclusion are also not chronic back pain, regular physical activity (3 or more times per week), women with pathological picture associated or malformation of the pelvic organs (secondary dysmenorrhea), or those that make use of device Intra- uterus (IUD).
* Will be excluded from the sample participants who submit two consecutive absences to care.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Estimated)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pain, Visual analog scale | two months
  Effects of pilates method in pain
Quality of health, score Short Form-36 | two months
  Effects of pilates method in quality of health

SECONDARY OUTCOMES:
Flexibility, finger-ground test | two months
  Effects of pilates method in flexibility

CONTACTS AND LOCATIONS:
Overall Officials: Juliany M A da Fonseca, Principal, Principal Investigator — Universidade Estadual do PiauÍ
Locations (1):
- Universidade Estadual do Piaui, Teresina, Piauí, Brazil